CLINICAL TRIAL: NCT01512680
Title: Evaluation of Functional Insulin Therapy on Blood Glucose Control in Type 1 Diabetic Patients Treated by Insulin Pumps
Brief Title: Evaluation of Functional Insulin Therapy in Type 1 Diabetic Patients
Acronym: IFOPI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 8749; ID-RCB : 2011-A00645-36 (Other: Afssaps)
Record Dates: First submitted 2011-12-16; First posted 2012-01-19 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Type 1 Diabetes
Keywords: Functional Insulin Thearpy; Carbs counting; Type 1 diabetes mellitus; Insulin pump; Treatment by external insulin pump
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Type 1 diabetes patient (Experimental): Type 1 diabetes patient are included in this study to have an education to Functional Insulin Therapy (intervention)
  Interventions: Behavioral: Education to Functional Insulin Therapy

INTERVENTIONS:
Behavioral: Education to Functional Insulin Therapy — * Intake of Continuous Glucose Monitor for 5 to 7 days
  * "Functional Insulinotherapy" training during 3 days, blood sampling, autoevaluation and QOL questionnary.
  * 1 month after the training: Follow-up consultation, clinical exam, vital signs and data on diabetes
  * 3 months after the training: Blood sampling, vital signs and data on diabetes
  * 6 months after the training: 2 sessions of training, blood sampling, autoevaluation and QOL questionnary, vital signs and data on diabetes, Intake of Continuous Glucose Monitor for 5 to 7 days
  * 9 months after the training: Blood sampling, vital signs and data on diabetes
  * 1 to 3 weeks before last visit: Intake of Continuous Glucose Monitor for 5 to 7 days
  * 12 months after the training: Follow-up consultation, clinical exam, vital signs and data on diabetes, autoevaluation and QOL questionnary

SUMMARY:
Functional Insulin Therapy (FIT) is an heath care method proposed to type 1 diabetic patients which focuses on patient autonomy, carbs counting and insulin dose adaptation. The hypothesis is that FIT should lead to better glycemic control (HbA1c), less hypoglycemia and better quality of life. 60 patient will be enrolled and followed during one year.

DETAILED DESCRIPTION:
Functional Insulin Therapy (FIT) is an heath care method proposed to type 1 diabetic patients which focuses on patient autonomy, carbs counting and insulin dose adaptation. In this study we plan to enroll 60 patients who will be educated toFIT and followed during one year. Patient will follow normal path of eductation which is composed of a 3 days inpatient admission, a medical visit one month after the education, and a 4hours reminder session six months after the education. We will compare HbA1c, hypoglycemia, weight, before the education, and after. Patient will also wear a continuous glucose sensor during one week before, at month 6 and month 12 to allow comparison of glucose variablity.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 70
2. Type 1 diabetes for more than 1 year
3. Treatment by basal/bolus insulin therapy and insulin pump for more than 6 months
4. HbA1c between 7.5 and 12%
5. Volunteer to be educated to Functional Insulin Therapy
6. Patient must be willing to undergo all study procedures
7. Patient must be affiliated or beneficiary of a social medical insurance
8. Patient has signed informed consent form prior to study entry

Exclusion Criteria:

1. Type 2 diabetes
2. Difficulties with mathematics calculation (simple algebra)
3. Patient is pregnant, or breast feeding during the period of the study
4. Manifest psychological disorders
5. Patient with eating behaviour desorder
6. Alcohol or drug addiction, as identified by investigator during screening visit
7. Persons deprived of freedom, adults protected by law or vulnerable persons

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2011-11; Primary Completion 2014-12 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Difference between HbA1c at Month 12 and Month 0 > 0.5% | at baseline et at Month 12

SECONDARY OUTCOMES:
Difference between HbA1c at Month 3 and Month 0 > 0.3% | at baseline et at Month 3
Difference between HbA1c at Month 6 and Month 0 > 0.5% | at baseline and at Month 6
Difference between HbA1c at Month 9 and Month 0 > 0.5% | at baseline and at Month 9
Reduction of 50% of hypoglycemia < 60mg/dl | at Month 12
Reduction of 30% of hypoglycemia between 60 and 80mg/dl | at Month 12
Reduction of number of patients who have severe hypoglycemia | at MONTH 12
Better score at surveys of quality of life (SF-6D, DQOL) and auto-management | at baseline, at Month 6 and at Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Eric ER RENARD, MD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Montpellier University Hospital, Montpellier, France